CLINICAL TRIAL: NCT02423928
Title: A Phase I Clinical Trial of Combined Cryotherapy and Intra-tumoral Immunotherapy With Autologous Immature Dendritic Cells in Men With Castration Resistant Prostatic Cancer and Metastases to Lymph Nodes and/or Bone Pre or Post Chemotherapy
Brief Title: Phase I Clinical Trial of Cryoimmunotherapy Against Prostate Cancer
Acronym: CryoIT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alden Cancer Therapy II (Industry)
Collaborators: Haukeland University Hospital (Other); Norwegian Radium Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACT2001; 2014-001898-14 (EudraCT Number)
Record Dates: First submitted 2015-04-15; First posted 2015-04-22 (Estimated); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Prostate Cancer
Keywords: immunotherapy; cryoablation; prostate cancer; dendritic cell
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Cyclophosphamide; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cryoimmunotherapy (Experimental): Patients with castration resistant prostate cancer and imaging proven metastases will be treated by autologous dendritic cell based cryoimmunotherapy of the prostatic tumor tissue assisted by immunomodulation consisting of low-dose metronomic cyclophosphamide for all patients plus ipilimumab for the latter half of all patients.
  Update January 2019: The protocol was changed as approved by the Norwegian Medicines Agency and the Regional Ethical Committee in Western Norway for the 3 last patients of altogether 18 patients. Consequently, the 3 last patients received 200 mg i.v. of pembrolizumab (and no ipilimumab) post-CryoIT.
  Interventions: Biological: Dendritic cell based cryoimmunotherapy; Drug: Cyclophosphamide; Drug: ipilimumab

INTERVENTIONS:
Biological: Dendritic cell based cryoimmunotherapy — Autologous dendritic cells will be obtained following leukapheresis and cytokine induction and will be injected into cryoablated prostate cancer tissue under ultrasound guidance.
  Other Names: ACT2001
Drug: Cyclophosphamide — Low-dose cyclophosphamide will be given metronomically for the purpose of selective inhibition of T regulatory cells for 6 months following start of treatment.
  Other Names: Sendoxan
Drug: ipilimumab — The antibody and immune checkpoint inhibitor ipilimumab (Yervoy) will be given for the last 10 patients enrolled into the study in addition to cryoimmunotherapy and low-dose cyclophosphamide.
  Other Names: Yervoy

SUMMARY:
20 patients with invasive castration resistant prostate cancer and radiologically verified metastases will be enrolled into the Phase I Clinical Trial. The trial is a dendritic cell based immunotherapy. Autologous dendritic cells will be obtained by leukapheresis and elutriation and stimulation by cytokines. The induced dendritic cells will have to pass viability, immunophenotyping and sterility criteria and will be injected into a cryoablated region of the primary prostate cancer tumor. The treatment is supplemented by immunomodulatory regimens.

DETAILED DESCRIPTION:
The study treatment dendritic cells (ACT2001) will be injected into the prostate following prostatic cryoablation. It is speculated that antigen from the cryoablated cancer will be available in the vicinity of the cryoablation field immediately following the procedure. Autologous, immature dendritic cells are capable of internalizing antigen, migrating to the lymphatic system, and presenting antigenic epitopes to T lymphocytes. In this way, dendritic cells are capable of initiating a cell-mediated systemic immune response.

In concept, the cancer itself should provide a specific and potentially broad spectrum of cancer-related antigens. Regulatory T lymphocytes, which have been implicated in dampening or halting cell-mediated, antigen-specific immune responses, will be selectively depleted using a regimen of low-dose cyclophosphamide. Low-dose cyclophosphamide has been empirically shown to selectively deplete the number of circulating regulatory T cells. The second half of patients will in addition receive treatment with the the immune checkpoint inhibitor ipilimumab antibody as one additional measure to avoid cancer cell immune evasion.

Using this combination of therapies, it is thought that a clinically significant anti-cancer immune response might be elicited.

ELIGIBILITY:
Inclusion Criteria:

* CRPC (castration resistant prostate cancer) with imaging study proven metastasis beyond pelvic lymph nodes and chemotherapy finished more than three months earlier
* Must be ambulatory with an ECOG performance status of 0 or 1
* No contraindications for MRI (pacemaker, claustrophobia, metal splints)
* Must be able to undergo the surgical procedure under general or regional anesthesia (spinal or epidural)
* Must be at least 18 years of age
* Must have lab values as the following :

White Blood Cells ≥ 1.5 x 10^9/L Platelets ≥ 100 x 10^9/L Hemoglobin ≥ 9g/dL (≥ 5.6 mmol/L) Creatinine ≤ 140 umol/L Bilirubin < 20% above the upper limit of normal ASAT and ALAT ≤ 2.5 the upper limit of normal Albumin ≥ 2.5 g/L sPSA < 200 ng/mL

• Signed informed consent and expected cooperation of the patients for the treatment and follow up must be obtained and documented according to ICH/GCP, and national/local regulations

Exclusion Criteria:

* History of other prior malignancy, with the exception of curatively treated basal cell or squamous cell carcinoma of the skin or effectively treated malignancy that has been in remission for over 5 years and is highly likely to have been cured
* Treatment with any other investigational medicinal product (IMP) within 4 weeks prior to first administration of study drug
* Adverse reactions to vaccines such as anaphylaxis or other serious reactions
* History of immunodeficiency or autoimmune disease such as rheumatoid arthritis, systemic lupus erythematosus, sclerodermia, polymyositis-dermatomyositis, juvenile onset insulin-dependent diabetes, or a vasculitic syndrome
* Significant cardiac or other medical illness that would limit activity or survival, such as severe congestive heart failure, unstable angina, or serious cardiac arrhythmia
* Active infection requiring antibiotic therapy
* Known hypersensitivity to any of the components of the cell therapy product
* Patients who test positive for hepatitis B, hepatitis C or HIV (Human Immunodeficiency Virus)
* Any other ongoing anti-tumor treatment (including chemotherapy, immunotherapy, cytokines, interferons, protease inhibitors or gene therapy) administered. The use of of GnRH-agonist/antagonists with or without bicalutamide is acceptable with the exception of GnRH-agonist with or without bicalutamide started up to 6 months prior to inclusion
* Use of not permitted concomitant medication: chronic corticosteroids except for asthma inhalers / topical use any agent with a known effect on the immune system, unless it is being given at dose levels that are not immunesuppressive, e.g. prednisone at 10mg/day or less
* Any alternative and complementary drugs that may affect the immune system or be potentially harmful to patients participating in phase I studies
* Any reason why, in the opinion of the investigator, the patient should not participate

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2019-08-16 (Actual)

PRIMARY OUTCOMES:
Composite measure of the safety and toxicity profile, including definition of the Maximum Tolerated Dose. | 72 weeks
  Maximum dose dendritic cells administered was well tolerated by interim analysis of 13 patients with database lock September 15th 2017
Pembrolizumab tested to boost dendritic cell-based immunity of patients 16 to 18 (3 last recruited patients to the trial). | 52 weeks
  200 mg pembrolizumab i.v. post-CryoIT was well tolerated - effect is under evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Beisland, MD PhD, Principal Investigator — Bergen Health
Locations (1):
- Haukeland University Hospital Research Department, Bergen, Hordaland, Norway

IPD SHARING:
Plan to Share IPD: Yes
Abstract published at Annual Meeting AACR 2018 in Chicago:
  http://www.aacr.org/Meetings/Pages/MeetingDetail.aspx?EventItemID=136#.WzNomaczZaS
  Abstract (Online) published Annual Meeting ASCO 2018 in Chicago:
  http://abstracts.asco.org/214/AbstView_214_219341.html
Access Criteria: The clinical trial has recruited all 18 patients by January 2019 in order to complete the Phase I clinical trial and with planned database lock and evaluation from August 2019. The interim analyses with database lock September 2017 concludes with good safety data and with therapeutic effects based upon analyses of radiology (stabilized disease of 5 of 13 patients), circulating tumor cells and ultradeep TCR-seq of CDR3 beta-chain of PBMC lymphocytes.